CLINICAL TRIAL: NCT04299178
Title: Human Factors Validation Testing for Use of the Belluscura X-PLO2R™ Portable Oxygen Concentrator (POC) System
Brief Title: Usability Evaluation of a Portable Oxygen Concentrator
Status: Completed | Type: Observational
Sponsor: Belluscura LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: BELL_XPLO2R
Record Dates: First submitted 2020-03-05; First posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Supplemental Oxygen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: X-PLO2R POC — Portable Oxygen Concentrator (POC)

SUMMARY:
This study evaluates how well an individual can put together and use a Portable Oxygen Concentrator (POC) by following the instructions in the User Manual.

DETAILED DESCRIPTION:
The Belluscura X-PLO2R Portable Oxygen Concentrator (POC) is intended for the provision of supplemental oxygen to patients with chronic pulmonary diseases, such as Chronic Obstructive Pulmonary Disease (COPD), and for a patient requiring supplemental oxygen, as prescribed by a physician. The purpose of this study is to evaluate if the X-PLO2R POC can be used by the intended users without serious errors or problems for the intended use and under the expected use conditions. Specifically, the study is to evaluate if potential users of the device can correctly, safely and effectively set-up, activate and operate the X-PLO2R POC to receive the required supplemental oxygen; if the intended user can understand and apply the information contained in the Belluscura X-PLO2R Quick Start Guide and User Manual; and to identify any and all use difficulties, problems and errors made during device assembly and operation, and to subsequently mitigate each identified instance of use error through device and/or materials modification, and to subsequently evaluate the effectiveness of each modification.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Male or female.
* Suitable for supplemental oxygen use from a suitably qualified and licensed medical professional.
* Voluntarily signed subject consent form.

Exclusion Criteria:

* Company employee.
* Former human factors study participants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population It is patients requiring supplemental oxygen, as prescribed by a physician.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Ability to correctly assemble and use the X-PLO2R POC | 2 hours
  A subject who is able to follow the instructions to correctly assemble and receive oxygen through the X-PLO2R POC will be considered a study pass.A subject who is not able to follow the instructions and does not correctly assemble and receive oxygen through the X-PLO2R POC will be considered a study fail.

CONTACTS AND LOCATIONS:
Overall Officials: Elvira Cawthon, MS, Principal Investigator
Locations (1):
- Belluscura LLC, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No